CLINICAL TRIAL: NCT03191305
Title: Comparison of the Efficacy of Rivroxaban to Coumadin( Warfarin ) in Cerebral Venous Thrombosis
Acronym: CVT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Foundation University Islamabad (Other)
Collaborators: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FUI/CTR/2017/2
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Cerebral Venous Thrombosis
MeSH Terms: conditions — Intracranial Thrombosis | interventions — Warfarin

STUDY DESIGN:
Intervention Model Description: Patients of CVT from Fauji Foundation would be be in Coumadin Arm ,and patients of CVT from Pakistan Institute of Medical Sciences Hospital would be in Rivroxaban arm.
Who Masked: Participant
Masking Description: Only Participants would not know about the any other choice of the Drug available.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coumadin Group (Active Comparator): Patients in Coumadin Group would be administered Coumadin with overlap of heparin for first two days followed by Coumadin given orally ,dose being adjusted according to INR .The INR range would be between 2-3.it would be given once a day.The total duration OFf coumadin would be six months.
  Interventions: Drug: Coumadin
- Rivoroxaban Group (Active Comparator): The dose protocol would be similar to the one used in Deep Venous Thrombosis. 15 mg PO q12hr for 21 days with food, THEN 20 mg PO qDay for 6 months.
  Interventions: Drug: Rivoroxaban

INTERVENTIONS:
Drug: Coumadin — Patients in Coumadin Group would be administered Coumadin with overlap of heparin for first two days followed by Coumadin given orally ,dose being adjusted according to INR .The INR range would be between 2-3.it would be given once a day. The total duration Of coumadin would be six months.
  Arms: Coumadin Group
Drug: Rivoroxaban — The dose protocol would be similar to the one used in Deep Venous Thrombosis. 15 mg PO q12hr for 21 days with food, Then 20 mg PO qDay for 6 months.
  Arms: Rivoroxaban Group

SUMMARY:
In past few years new anticoagulants have been developed which directly inhibit thrombin or factor X.factor x inhibitor is available in Pakistan. The superior efficacy of Rivroxaban has been shown in Deep Venous Thrombosis in EINSTEIN study (3).Its definite superiority in prevention of embolic stroke in nonvalvular atrial fibrillation is evidenced by the study ROCKET AF (4). With Rivroxaban no monitoring is required, and also there are no drug interactions .There are few pilot studies of using Rivroxaban in cerebral venous thrombosis. This study is therefore required to find its efficacy in CVT patients as well as its comparison with Coumadin

DETAILED DESCRIPTION:
Cerebral venous thrombosis is rare form of stroke, accounting .5 to 1% only (1)Exact estimate for Pakistani population is not known Mubarak et al described 6- year imaging incidence and prevalence of CVST to be 10.22% and 11.055% respectively(2) .Majority of cerebral venous stroke patients are females in reproductive age. Coumadin is one of the notorious drugs to be used in pregnancy categorized as X. it also has many drug interactions .and there are diet restrictions too being on Coumadin. It also requires maintanence of prothrombin time in certain range which means patient has to go under phlebotomy at least twice a month. Moreover not all laboratories are well equipped resulting in poor test sensitivity. and at times clinicians keep patients on suboptimum doses for fear of bleeding ending with poor efficacy.

In past few years new anticoagulants have been developed which directly inhibit thrombin or factor X.factor x inhibitor is available in Pakistan.

The superior efficacy of Rivroxaban has been shown in Deep Venous Thrombosis in EINSTEIN study (3).Its definite superiority in prevention of embolic stroke in nonvalvular atrial fibrillation is evidenced by the study ROCKET AF (4). With Rivroxaban no monitoring is required, and also there are no drug interactions .There are few pilot studies of using Rivroxaban in cerebral venous thrombosis. This study is therefore required to find its efficacy in CVT patients as well as its comparison with Coumadin .

OBJECTIVE To Compare the efficacy of Rivroxaban to Warfarin in Cerebral Venous Thrombosis MATERIAL AND METHODS STUDY DESIGN: Quasi Experimental; Descriptive cross sectional

DURATION OF STUDY:

6 months to 1 year

SAMLE SIZE :

50 patients SAMPLING TECHNIQUE : Consecutive (non probability) sampling.

INCLUSION CRITERIA:

Patients of either gender Age between 13 years and 50 years Patients with proven CVT on neuro imaging (CTV, o MRV)

EXCLUSION CRITERIA:

Patients suffering from Chronic Liver disesase Patients having contraindications for oral anticoagulation Patients suffering from hematological or brain malignancy Patients whose MRV and CTV do not support CVT

DATA COLLECTION PROCEDURE After taking permission from hospital ethical review committee , All patients with confirmed CVT based on established criteria using any NOAC or WARFARIN presenting to PIMS or FFH hospitals will be enrolled. Data will be obtained by retrospective manner if they are using anticoagulants for more than 6 months. If patients are using anticoagulants for less than 6 months, they will be enrolled and followed up for six months.

DATA ANALYSIS The data will be analyzed using SPSS version 16.0. Descriptive analysis will be done and reported as mean ± SD for continuous variables like age whereas frequencies and percentages will be calculated for categorical variables such as gender, individual risk factors.

P-value ≤ 0.05 will be significant. Results will be presented in tabulated or graphical forms.

Outcome measures Outcome measures will include any hemorrhage or recurrent CVT based on repeat MRI.

MRs Scale Secondary Outcome Comparison of cost of two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

Patients of either gender Age between 13 years and 50 years Patients with proven CVT on neuro imaging (CTV, o MRV) -

Exclusion Criteria:

Patients suffering from Chronic Liver disesase Patients having contraindications for oral anticoagulation Patients suffering from hematological or brain malignancy Patients whose MRV and CTV do not support CVT

-

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Hemorrhage or Recurrent CVT based on repeat MRI. | 6 months
  Outcome measures will include any hemorrhage or recurrent CVT based on repeat MRI.

SECONDARY OUTCOMES:
Cost | 6 months
  Comparison of cost of two treatment groups.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stam J. Thrombosis of the cerebral veins and sinuses. N Engl J Med. 2005 Apr 28;352(17):1791-8. doi: 10.1056/NEJMra042354. No abstract available. PMID 15858188
- [Background] F. Mubarak, A. Muhammad, Cerebral venous sinus thrombosis: Incidence, prevalence and patterns of neurological involvement: a retrospective study from Pakistani population European society of Radiology .
- [Background] EINSTEIN Investigators; Bauersachs R, Berkowitz SD, Brenner B, Buller HR, Decousus H, Gallus AS, Lensing AW, Misselwitz F, Prins MH, Raskob GE, Segers A, Verhamme P, Wells P, Agnelli G, Bounameaux H, Cohen A, Davidson BL, Piovella F, Schellong S. Oral rivaroxaban for symptomatic venous thromboembolism. N Engl J Med. 2010 Dec 23;363(26):2499-510. doi: 10.1056/NEJMoa1007903. Epub 2010 Dec 3. PMID 21128814
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Background] Anticoli S, Pezzella FR, Scifoni G, et al. Treatment of Cerebral Venous Thrombosis with Rivaroxaban. J Biomedical Sci.